CLINICAL TRIAL: NCT02328040
Title: Double-blinded, Randomized, Controlled Paired Trial Comparing Sitagliptin to Placebo in Closed Loop.
Brief Title: Randomized Trial Comparing Sitagliptin to Placebo in Closed Loop
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Rubina Heptulla, Division Chief of Pediatric Endocrinology, Albert Einstein College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-330-000
Record Dates: First submitted 2014-09-11; First posted 2014-12-31 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Closed loop; Artificial Pancreas; Insulin; Sitagliptin; Januvia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Sitagliptin Phosphate; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Placebo Comparator): Placebo and Insulin monotherapy via CL
  Interventions: Drug: Placebo and Insulin monotherapy via CL
- Part B (Active Comparator): Sitagliptin and insulin/novolog via CL
  Interventions: Drug: Sitagliptin and insulin/novolog via CL

INTERVENTIONS:
Drug: Placebo and Insulin monotherapy via CL — In the control arm patient receives a placebo pill with the closed loop with insulin/novolog (placebo and insulin/novolog via CL)
  Arms: Part A
Drug: Sitagliptin and insulin/novolog via CL — In the treatment arm the participant receives a single dose of sitagliptin with closed loop with insulin/novolog (Sitagliptin and insulin/novolog via CL), Part B
  Other Names: Januvia
  Arms: Part B

SUMMARY:
There are many recent advances in insulin treatment of type 1 Diabetes Mellitus (T1DM), however after a meal sugars are always a concern. There is a drug sitagliptin (Januvia) which is FDA approved to treat people with type 2 diabetes which helps correct their glucose (sugars) after meals. This study is going to test whether this drug can improve the after meal sugars in people with type 1 diabetes. To test this, you will be given a mixed meal and its effects on insulin levels. The hormones that affect blood glucose as well as your sugar levels will be measured by a series of blood tests. We will also look for high blood sugars which might occur because of food staying longer in the stomach than usual or due to the suppression of a hormone called glucagon which increases blood sugar. If you qualify, you will be given sitagliptin (Januvia) 50 mg and 100 mg dosages. You and the researchers will not know which dose you are taking at any single visit. We will first enroll 10 subjects with established type 1 Diabetes Mellitus for at least 1 year, between the ages of 18-30 years old. The first 10 patients will be evaluated for safety parameters such as ability to keep blood sugars < 70 mg/dl for at least 70% of the time, no episode of severe hypoglycemia (low blood sugars) and so on. After this safety criteria is established, we will then recruit subjects between the ages of 14-19 yrs for the next phase of the study. A total of 17 subjects were enrolled into the study.

DETAILED DESCRIPTION:
Rationale: Sitagliptin has been extensively studied in patients with type 2 Diabetes Mellitus (T2DM). Sitagliptin increases endogenous GLP-1 (Glucagon like peptide) by inhibiting the break down of an enzyme DPP-4 (Dipeptidyl Peptidase 4). GLP-1 in turn results in glucagon suppression.This mechanism is very effective in improving after meal blood sugars, not only in type 2 diabetics but also in type 1 diabetes. In this study we will test the use of sitagliptin in decreasing after meal blood sugars in the setting of closed loop.Data Safety Monitoring Board (DSMB) will meet before the initiation of the study and before children are enrolled into the study. The safety data after the meeting will be submitted to the Institutional Review Board (IRB).

Specific Aim: In the closed loop setting, to establish a safe and an effective dose of sitagliptin in type 1 diabetes (T1DM) compared to placebo and its effects in lowering the post meal glucose levels, Further to test its effects on insulin utilization , glucagon levels and gastric emptying.

Hypothesis: Post meal sugars will decrease in a dose dependent manner due to glucagon suppression when sitagliptin is used in the closed loop setting as compared to placebo.

Study Design: Following informed consent (and with appropriate subject assent), each subject with Type 1 DM will undergo 4 study visits: Screening , Part A (Placebo/Insulin) and Part B (Sitagliptin 100 mg). A randomized double-blinded 2-period cross over study trial will be used for the subjects to participate in the study . All the study subject's (18-30 yrs old) and the study staff (except one person) will be blinded to the study parts and they will do all the study Parts A and B in random order.

Montefiore Medical Center (MMC) Investigational pharmacy and one of the study staff (excluding the PI) will be un-blinded to the protocol for doing the randomization table, dispensing, checking the dose of study medication and scheduling the study visits (done by the study staff person). The participants will be admitted to the Clinical Research Center (CRC) on two occasions for the Parts A and B following the screening visit. Parts A and B are done with at least 2 weeks apart.

Inclusion/ Exclusion Criteria: Subjects with Type 1 DM in the age group of 14-35 years without any concomitant illnesses except treated hypothyroidism will be recruited and also have an HbA1C less than 8.5 %. Menstruating women must have a negative pregnancy test. Lactating and pregnant women will be excluded and anyone with anemia defined by Hemoglobin of less than 12 gm/dl. Also, subjects with a history of substance abuse (evaluated by medical history and CRAAFT questionnaire which will be administered at the screening visit) will be excluded. The subject's should not be on any other medication which affects blood sugars.

Screening: After signing a consent form, a screening evaluation will be performed 4-6 weeks prior to study enrollment in the CRC. The evaluation will consist of medical history, physical examination (including height, weight, vital signs and tanner staging), and blood samples for clinical laboratory tests: CBC (complete blood count), Liver Function Tests (LFT's), amylase, lipase, creatinine and HemoglobinA1C (HbA1C). The approximate volume of blood drawn is expected to be 12 ml. CRAAFT questionnaire will be administered. Subjects will undergo a baseline blinded open loop evaluation using a Medtronic CGM iPro 2 (Continuous Glucose Monitoring System) which is the insertion device. It has three parts - a glucose sensor that is inserted subcutaneously, a transmitter which connects to the sensor electrode and is attached to the body and a receiver which displays the glucose values.

Part A: The subjects will be admitted to the Clinical Research Center (CRC) around 2 PM on day 1. Vitals will be taken. IV will be placed and blood will be drawn to measure Stat CBC, HbA1C, Liver function tests, Serum Amylase, Serum Lipase and Serum Creatinine. Study will be continued only if their Hemoglobin is greater than 12 gm/ dl. Urine pregnancy test will be done for all female subjects prior to study. Insulin infusion through the subcutaneous pump will be continued or long acting analog, novolog will be given as per home regimen. Subjects will be on the continuous glucose monitoring system overnight till 9 PM on day 2.

BLOOD SAMPLING AND MEDICATIONS: At 6.30 PM on day 1 subjects will be started on the closed-loop device for the automated delivery of insulin based on the glucose sensor measurements . The insulin dose will be based on the patient's usual insulin to carbohydrate ratio. Placebo pill will be given around 8 PM (0 min) and then dinner will be served as a carbohydrate consistent diet (60 gms of carbohydrate). Subjects will be on the closed loop device over night till 9 PM on day 2. On day 2 breakfast will be served at 7 AM (660 min) in the morning consisting of a boost (high protein drink) 9.6 oz, consumed over a period of 10-15 min. Lunch and dinner will be served at 12 PM (960 min) and 5 PM (1260 min). At approximately 6.30 PM baseline blood samples will be drawn prior to study start for glucose, insulin, glucagon, GLP-1, DPP-4 activity and Sitagliptin. Also, there will be blood draws at the following time points: 0, 60, 120, 240, 360, 480, 540, 600, 660, 720, 780, 840, 900, 960, 1020, 1080, 1140, 1200, 1260, 1320, 1380, 1440. The insulin pump basal rate (or novolog) will be set to continue as per home regimen. Blood glucose concentrations will be measured at the bedside using an Analox glucose analyzer. The subject will be discharged after this. They will not be paid separately for transportation, parking or child care. A social security number will be required. It will be kept confidential. For minors, compensation will be given to the parent, but it is intended for the child.

A subject will be withdrawn from participating in the study if he/she meets any of the following conditions: 1) develops a chronic disease 2) develops anemia 3) becomes pregnant 4) develops a weight loss of greater than 10 pounds for unspecified reasons 5) loss of contact- if we are unable to reach a study subject (within 2 months of screening or completion of the first study) by phone or mail to schedule the next appointment. All study subjects (that are withdrawn from the study) will receive a phone call and a letter notifying them that they have been withdrawn. Blood samples will be kept for 20 years because some of the assays have not been developed for some of the hormone analyses. Since it is difficult to perform clinical studies in pediatrics, we feel it is better to bank blood samples and perform hormone analyses as newer assays become available rather than repeating the study.

Part B: Will be identical as part A except that Sitagliptin 100 mg will be administered as a pill before dinner at 8 PM on day 1. In Part B urine pregnancy test will be done before the visit for all female subjects. Prior to each part, hemoglobin must be >12 g/dl and a female subject should test negative for pregnancy.

Treatment of Hypoglycemia: If blood glucose values in a subject are less than 55 mg/dl, IV glucose of 5-10gm, or if blood glucose less than 50 mg/dl, 10-15 g will be administered for countering low blood glucose to achieve euglycemia (90-130 mg/dl). 1-2 doses of IV glucose should correct hypoglycemia. If more than 3-4 doses are required to achieve euglycemia, the study will be terminated and the subjects will be offered a meal tray and blood sugar rechecked to ensure euglycemia. After the completion of the first 2 study subjects, the data safety and monitoring committee will assess safety of the protocol, as well as drug doses and adjustments to the protocol will be made. If hypoglycemia occurs even with the reduced dose of insulin, further reduction in insulin dose will be advised. The total blood draw volume will be 95 cc (1/2 cup) for Part A and B.

Statistical Analysis :

Sample size: Data from an earlier trial determined that the mean area under the curve (AUC) for children with Type 1 DM with insulin alone was 470 mg*hr/dl. The current trial is designed to detect a 25% difference in mean area under curve (AUC) for glucose in the 1670 min period. Based on power of 0.8, alpha of 0.05 and correlation coefficient of r >/= 0.5 (based on previous studies) and standard deviation excursion measure AUC for glucose approximately 0.8 between two study conditions, we estimate a sample size of 16 subjects. With a usual 10% drop out rate noticed in our studies , we would need to recruit 17 subjects.

Data Analysis: Two way analysis of variance (ANOVA) for repeated measures will be used to compare between the two study periods, insulin , glucagon and glucose concentrations over time. Mean area under the curve (AUC) over the time will be calculated and a modified paired t-test will be used for post hoc analysis.Differences will be considered significant at 0.05. Comparative and descriptive statistics will be computed using SPSS (Statistical Package for the Social Sciences) statistical software and Graph pad prism.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 14 to 30 years
2. Subjects must be otherwise healthy except for T1DM, and treated for hypothyroidism if present
3. Menstruating women must have negative pregnancy test.
4. Hemoglobin (Hb) more than 12 g/dl

Exclusion Criteria:

1. Having any other chronic condition except hypothyroidism stable on medications
2. On chronic medications that may affect glucose excursions
3. Hemoglobin less than 12 g/dl
4. Positive pregnancy test (based on Urine)
5. Pregnant or lactating mothers Known allergy to Januvia-

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Heptulla, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine CRC, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 participants were screened. However, only 17 participants were enrolled and of these 15 participants completed both study visits. Patients were recruited from diabetes clinics, via fliers, and online postings on clinical trial sites.
Groups:
- Placebo/Insulin First, Then Sitagliptin/Insulin: Participants first received Placebo/Insulin, placebo orally and Insulin subcutaneously for 2 days. Then they received Sitagliptin/Insulin, 100 mg of Sitagliptin orally and insulin subcutaneously for the next 2 days. Each visit is 3-4 weeks apart.
- Sitagliptin/Insulin First, Then Placebo/Insulin: Participants first received Sitagliptin/Insulin, 100 mg of Sitagliptin orally and insulin subcutaneously for the next 2 days. Then they received Placebo/Insulin, placebo orally and Insulin subcutaneously for the next 2 days. Each visit is 3-4 weeks apart.
Period: First Intervention (2 Days)
Arm/Group | Placebo/Insulin First, Then Sitagliptin/Insulin | Sitagliptin/Insulin First, Then Placebo/Insulin
Started | 8 | 9
Completed | 7 | 8
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention (2 Days)
Arm/Group | Placebo/Insulin First, Then Sitagliptin/Insulin | Sitagliptin/Insulin First, Then Placebo/Insulin
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Placebo/Insulin Participants, placebo orally and Insulin subcutaneously or Sitagliptin/Insulin, 100 mg of Sitagliptin orally and insulin subcutaneously.
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Measures in Subjects Treated With Sitagliptin, Compared to the Placebo
Description: Better targeted blood glucose levels in the CL setting in the treatment arm, Sitagliptin, compared to placebo (insulin monotherapy)
Time Frame: 18 Months
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Placebo/Insulin: Participants who received Placebo/Insulin, placebo orally and Insulin subcutaneously for 2 days.
- Sitagliptin/Insulin: Participants who received Sitagliptin/Insulin, 100 mg of Sitagliptin orally and insulin subcutaneously for 2 days.
Arm/Group | Placebo/Insulin | Sitagliptin/Insulin
Number analyzed (Participants) | 15 | 15
mg/dl | 149.7 (37.8) | 155.9 (48.6)

2. Secondary Outcome: Measure of Glucagon Concentration in Subjects Treated With Sitagliptin, Compared to Placebo
Description: Serum glucagon concentrations were measured in the CL setting in the treatment arm, sitagliptin, compared to the placebo (Insulin monotherapy)
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: Pmol/L
Arm/Group | Placebo/Insulin | Sitagliptin/Insulin
Number analyzed (Participants) | 15 | 15
Pmol/L | 6.04 (1.5) | 5.66 (1.6)

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Siatagliptin/Insulin: Participants who received Sitagliptin/Insulin, 100 mg of Sitagliptin orally and insulin subcutaneously for 2 days.
Arm/Group | Placebo/Insulin | Siatagliptin/Insulin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No